CLINICAL TRIAL: NCT03756649
Title: Mayo Clinic IBD Biobank
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 18-007941
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; Ulcerative colitis; Crohn's
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood work to be obtained from patient to be processed and stored until needed in the future for potential research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Subjects without inflammatory bowel disease (IBD) will have samples collected of blood, urine and stool
  Interventions: Procedure: Blood Draw; Procedure: Urine Collection; Procedure: Stool Collection
- Inflammatory bowel disease (IBD): Subjects with known inflammatory bowel disease will have samples collected of blood, urine and stool
  Interventions: Procedure: Blood Draw; Procedure: Urine Collection; Procedure: Stool Collection

INTERVENTIONS:
Procedure: Blood Draw — 50 ml will be collected
Procedure: Urine Collection — 50 ml will be collected
Procedure: Stool Collection — Three 25 ml tubes will be collected

SUMMARY:
Researchers are collecting and storing blood, stool, and urine samples and medical information to better understand Inflammatory Bowel Disease (IBD) to improve disease outcome.

DETAILED DESCRIPTION:
Subjects will be sent a letter detailing the proposed biobank and soliciting enrollment. Following the informed consent process, subjects will provide a blood sample (50 ml), urine sample (50 ml), and stool. The blood and urine samples will either be collected at the one of the Mayo Clinic outpatient laboratories or by a mail-out kit. Subjects will be asked to complete a questionnaire and 24-hour food recall questionnaire (completed online).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with inflammatory bowel disease (IBD) who are between the ages of 18 and 85 at time of study enrollment.
* The diagnosis of IBD will be based on the standard IBD criteria including biochemical and colonoscopy screening.
* Women with inflammatory bowel disease of childbearing potential and pregnant women will be offered enrollment because there is no risk to an unborn child in this investigation.
* Patients between the ages of 18 and 85 without history of IBD or colon cancer.

Exclusion Criteria:

* Patients with known liver disease.
* Patients unable to provide informed consent.
* Prisoners and institutionalized individuals.
* Patients with a history of colorectal cancer.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with inflammatory bowel disease (IBD) who are between the ages of 18 and 85 at time of study enrollment.
  * The diagnosis of IBD will be based on the standard IBD criteria including biochemical and colonoscopy screening.
  * Women with inflammatory bowel disease of childbearing potential and pregnant women will be offered enrollment because there is no risk to an unborn child in this investigation.
  * Patients between the ages of 18 and 85 without history of IBD or colon cancer.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2065-12 (Estimated); Study Completion 2065-12 (Estimated)

PRIMARY OUTCOMES:
Study Participants | 50 years
  Total number of participants in the study

SECONDARY OUTCOMES:
Urine Collection | 50 years
  Total number of urine samples collected
Blood Collection | 50 years
  Total number of blood samples collected
Stool Collection | 50 years
  Total number of stool samples collected

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N. Lazaridis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States